CLINICAL TRIAL: NCT06561542
Title: A Phase I, Escalating Single and Multiple Dose Study of LX22001 for Injection to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Bioavailability in Healthy Subjects.
Brief Title: A Phase I Study of LX22001 for Injection in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NE862401
Record Dates: First submitted 2024-08-06; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — tegoprazan; Esomeprazole; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LX22001 for Injecton (Experimental)
  Interventions: Drug: LX22001 for Injeciton
- Tegoprazan tablet (Active Comparator)
  Interventions: Drug: Tegoprazan tablet
- Esomeprazole sodium for injection (Active Comparator)
  Interventions: Drug: Esomeprazole sodium for injection

INTERVENTIONS:
Drug: LX22001 for Injeciton — single dose: 25mg,50mg,100mg,200mg ,intravenous infusion. repeat doses: 50mg,100mg , intravenous infusion,once daily for 3 days.
  Arms: LX22001 for Injecton
Drug: Tegoprazan tablet — 50mg,oral,single dose
  Arms: Tegoprazan tablet
Drug: Esomeprazole sodium for injection — 80 mg intravenous infusion for 30 min followed by a continuous infusion of 8 mg/h for 71.5h
  Arms: Esomeprazole sodium for injection

SUMMARY:
Study to evaluate the safety and tolerability, pharmacokinetics/pharmacodynamics (PK/PD) parameters of an escalating, single dose/repeat doses of LX22001 for injection in healthy subjects.

ELIGIBILITY:
"Inclusion Criteria:

1. Subjects who fully understand the objectives, nature, methods and possible AEs of the study, voluntarily participate in the clinical study, and sign the Informed Consent Form (ICF) before the initiation of any study procedure, and warrant that any study procedure will be participated in by themselves;
2. Healthy Chinese subjects aged 18-45 years (inclusive, at the date of signing the ICF), both males and females;
3. Body mass index (BMI): 19.0-26.0 kg/m2 (inclusive); weight: ≥ 50 kg for male and ≥ 45 kg for female;
4. Subjects who are willing to use effective contraception and have no sperm or egg donation plan from the time of signing the informed consent form until 3 months after the last dose (see Appendix 20.1 for details of contraceptive measures and contraceptive requirements);
5. Subjects who can communicate well with the investigator, and understand and comply with the requirements of this study."

"Exclusion Criteria:

1. Allergy (such as: allergic to two or more drugs, foods, or pollen), history of atopic allergic disease (such as: asthma, urticaria, eczematous dermatitis, etc.), history of allergy to any of the components and excipients of the study drugs (LX22001 for injection, tegoprazan tablets, and Esomeprazole Sodium for injection), or allergy to penicillin, cephalosporin, and other antibiotics;
2. Any disease or history of disease that may significantly affect drug absorption, distribution, metabolism, and excretion, or any condition that may pose a hazard to the subject, such as: inflammatory bowel disease, gastric ulcer, duodenal ulcer, gastrointestinal/rectal bleeding, persistent nausea, or other clinically significant gastrointestinal anomalies; history of major gastrointestinal surgery (such as: gastrectomy, gastrointestinal anastomosis, bowel resection, gastric bypass, gastric banding, cholecystectomy, except for appendicitis surgery and prolapse surgery);
3. History of chronic or serious illness or present illness of cardiovascular, hepatic, renal, respiratory, hematologic and lymphatic, endocrine, immunologic, psychiatric, neurologic, gastrointestinal, metabolic, and skeletal systems within the last 1 year;
4. Clinically significant abnormalities in physical examination and laboratory tests at screening, judged by the investigators;
5. For those with clinically significant abnormalities in vital signs at screening which will be judged by the investigators based on the actual situations;
6. The serological virology test shows positive results of HIV antigen antibody (HIV-Ag/Ab), hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), or treponema pallidum antibody (TP-Ab) at screening;
7. Women who have not taken effective contraception within 15 days prior to the screening period, or have a positive blood pregnancy test or are breastfeeding during the screening period;
8. Those who have a history of drug abuse within the past five years or drug use in the three months prior to screening, or positive results for urine drug test during the screening period;
9. Those who smoke more than 5 cigarettes per day or had a habit of using nicotine-containing products within 3 months prior to screening, or test positive for nicotine test at screening;
10. Those who drink more than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of ABV 40% spirit or 150 mL of wine) within 3 months prior to screening or have consumed an alcohol-containing product 48h prior to the dose or test positive for alcohol breath test at screening;
11. Those who have used any medication (including prescription, over-the-counter, nutritional supplements, Chinese herbal medicine, vitamins, etc.) or are on medication within 1 month prior to screening;
12. Those who have participated in other clinical studies and used other investigational drugs or interventional therapies within 3 months prior to screening;
13. Those who have donated or lost more than 200 mL of blood or received blood transfusion or used blood products within 3 months prior to screening;
14. Those who have consumed any food or beverage containing caffeine or producing caffeine or xanthine metabolites (e.g., coffee, tea, chocolate) within 48h prior to the dose;
15. Those who have consumed grapefruit, limes, carambola,pitaya, mango or food or drinks prepared from them within 7 days prior to screening;
16. Those who are unable to establish intravenous access or intolerable to intravenous administration;
17. Those who are involved in the planning and execution of this study;
18. Any other circumstance that, in the opinion of the investigator, the subject may be hindered from providing informed consent or following the protocol, or the subject's participation in the study may affect the results of the study or his or her own safety."

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 7 days from dosing

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to the 24-Hour Time Point (AUC0-24) | pre-dose to Day1 post-dose
Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) | pre-dose to Day1 post-dose
Maximum Observed Plasma Concentration (Cmax) | pre-dose to Day1 post-dose
Terminal elimination half-life(t1/2) | pre-dose to Day1 post-dose
Apparent total body clearance (CL) | pre-dose to Day1 post-dose
Apparent volume of distribution(Vd) | pre-dose to Day1 post-dose
Area Under the Concentration-Time Curve During a Dosing Interval (AUCtau) at Steady State | Day 3 post-dose
Cmax at Steady State (Cmax,ss) | Day 3 post-dose
Percentage of Time Gastric pH above 4 over 24h | baseline, Day 1 and Day 3
Percentage of Time Gastric pH above 6 over 24h | baseline, Day 1 and Day 3
Mean Gastric pH over 24h | baseline, Day 1 and Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Hongyun Wang, Principal Investigator — Peking Union Medical College; Hongzhong Liu, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China